CLINICAL TRIAL: NCT05108870
Title: A Randomized Phase I/II Trial of TheraT® Vectors Expressing HPV16 Specific Antigens in Combination With Neoadjuvant Chemotherapy Followed by Transoral Robotic Surgery or Risk/Response Stratified Chemoradiotherapy for Locoregional HPV16+ Oropharyngeal Cancer
Brief Title: TheraT® Vectors (Vaccines) Combined With Chemotherapy to Treat HPV16 Head and Neck Cancers
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IRB21-1031
Record Dates: First submitted 2021-10-25; First posted 2021-11-05 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Human Papilloma Virus; HPV; HPV Positive Oropharyngeal Squamous Cell Carcinoma; Head and Neck Cancer
Keywords: throat cancer; human papilloma virus; HPV16; head and neck cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1: Dose-Finding Group 1 - Drug Combination 1 (Experimental): All participants in this group will receive HB-201 combined with chemotherapy using carboplatin and paclitaxel.
  - HB-201 will be administered on cycle 1 day 15, cycle 2 day 15, and cycle 3 day 15 with three 21-day cycles of carboplatin on day 1 and paclitaxel 100mg/m2 on days 1, 8, and 15
  Interventions: Drug: HB-201; Drug: HB-202; Drug: Carboplatin; Drug: Paclitaxel
- Phase 1: Dose-Finding Group 2 - Drug Combination 2 (Experimental): All participants in this group will receive alternating doses of HB-201 and HB-202 combined with chemotherapy using carboplatin and paclitaxel.
  Participants will be given 3 doses of HB-201 & HB-202 alternating two vector therapy. Patients will receive 2 doses of HB-202 and 1 dose of HB-201. HB-202 will be administered on cycle 1 day 15 and cycle 3 day 15, and HB-201 will be administered on cycle 2 day 15 with three 21-day cycles of chemotherapy with carboplatin on day 1 and paclitaxel 100mg/m2 on days 1, 8, and 15.
  Interventions: Drug: HB-201; Drug: HB-202; Drug: Carboplatin; Drug: Paclitaxel
- Phase 2: Efficacy Arm 1 - HB-201 + Chemotherapy (Experimental): Participants in this group will receive HB-201 combined with chemotherapy using carboplatin and paclitaxel at the dose established in the first phase of the study.
  After completing treatment at the established phase 2 dose, subjects will receive surgery, radiotherapy alone, or chemotherapy with radiotherapy together based on how their tumor responds to the medications.
  Interventions: Drug: HB-201; Drug: HB-202; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Transoral Robotic Surgery
- Phase 2: Efficacy Arm 2 - HB-201 and HB-202 + Chemotherapy (Experimental): Participants in this group will receive alternating doses of HB-201 and HB-202 combined with chemotherapy using carboplatin and paclitaxel at the dose established in the first phase of the study.
  After completing treatment at the established phase 2 dose, subjects will receive surgery, radiotherapy alone, or chemotherapy with radiotherapy together based on how their tumor responds to the medications.
  Interventions: Drug: HB-201; Drug: HB-202; Drug: Carboplatin; Drug: Paclitaxel; Procedure: Transoral Robotic Surgery

INTERVENTIONS:
Drug: HB-201 — A anti-cancer vaccine that treats HPV-related cancers.
  Other Names: TheraT® Vectors
Drug: HB-202 — A anti-cancer vaccine that treats HPV-related cancers.
  Other Names: TheraT® Vectors
Drug: Carboplatin — Chemotherapy drug.
Drug: Paclitaxel — Chemotherapy drug.
Procedure: Transoral Robotic Surgery — Transoral robotic surgery is a procedure to remove mouth and throat cancers in which a surgeon uses a sophisticated, computer-enhanced system to guide the surgical tools.
  Other Names: TORS
  Arms: Phase 2: Efficacy Arm 1 - HB-201 + Chemotherapy; Phase 2: Efficacy Arm 2 - HB-201 and HB-202 + Chemotherapy

SUMMARY:
Doctors leading this study hope to learn about the safety and effectiveness of combining medications HB-201 and HB-202 (also known as TheraT® vectors) with chemotherapy using carboplatin and paclitaxel in the beginning of the study (induction) and if combining these medications can increase tumor shrinkage after therapy and reduce the amount of radiotherapy and chemotherapy that will later be needed.

In addition, the study is looking at ways to reduce side effects overall using robotic surgery, chemotherapy and radiotherapy, or radiotherapy alone. Your participation in this research will last about 2 years.

HB-201 and HB-202 are experimental (meaning the US Food and Drug Administration (FDA) has not approved these drugs), and therefore they can only be given in a research study.

ELIGIBILITY:
INCLUSION CRITERIA

1. Subjects must have clinically confirmed human papilloma virus (HPV)16-positive head and neck squamous cell carcinoma of the oropharynx. Confirmed HPV-positive disease of other subsites are uncommon but also eligible.
2. Must have HPV16 subtype demonstrated based on clinical guidelines established by the study doctor.
3. Availability of ≥10 unstained 5 micron slides (to be provided to Human Tissue Resource Center at the University of Chicago). Participants who cannot fulfill this requirement will need to undergo a new biopsy prior to enrollment on study.
4. Participants must be at least 18 years of age.
5. Subjects with American Joint Committee on Cancer (8th edition, 2018) N1 (solitary lymph node >=3cm), N2-N3 nodal disease or T3-T4 primary tumor (with any N).
6. Measurable disease (either primary site and/or nodal disease) by Response Evaluation Criteria in Solid Tumors 1.1.
7. No previous radiation or chemotherapy for a head and neck cancer.
8. No complete surgical resection for a head and neck cancer within 8 weeks of enrollment (although lymph node biopsy including excision of an individual node with presence of residual nodal disease, or surgical biopsy/excision of the tumor with residual measurable disease is acceptable.) No surgical procedures or biopsies will occur after baseline scans are performed and measurable lesions are identified.
9. Eastern Cooperative Oncology Group performance status 0-1
10. Normal Organ Function as confirmed by clinical lab values.
11. Must be considered to be a candidate to receive cisplatin by the treating physician.
12. Must sign a study-specific informed consent form prior to study entry. Patients should have the ability to understand and the willingness to sign a written informed consent document.
13. Women of childbearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 24 hours prior to the start of study drug.
14. Women must not be breastfeeding.
15. Women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment.
16. Men who are sexually active with women of childbearing potential must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s).

EXCLUSION CRITERIA

1. Unequivocal demonstration of distant metastatic disease (M1 disease).
2. Non-HPV16 subtype.
3. Unidentifiable primary site.
4. Intercurrent medical illnesses that impairs the patient's tolerance to therapy or limits survival. This includes but is not limited to ongoing or active infection, immunodeficiency, symptomatic congestive heart failure, pulmonary dysfunction, cardiomyopathy, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance. Patients with clinically stable and/or chronically managed medical illnesses that are not symptomatic and/or are not expected to impact treatment on protocol are still eligible (conditions to be reviewed by the PI to confirm eligibility).
5. Active, known, or suspected, autoimmune or inflammatory disorders requiring immunosuppressive therapy, with the exception of low-dose prednisone (<= 10mg or equivalent). The following are exceptions to these criteria:

   * Patients with vitiligo or alopecia.
   * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
   * Any chronic skin condition that does not require systemic treatment.
6. Treatment with any chronic immunosuppressive medication within six months prior to the first administration of study treatment (unless agreed otherwise).
7. Participants who have had a prior anaphylactic or other severe reaction to human immunoglobulin or antibody formulation administration.
8. Herbal remedies with immune-stimulating properties or known to potentially interfere with major organ function within 28 days prior to the first dose of study treatment, unless agreed otherwise with the primary investigator.
9. Prior surgical therapy other than incisional/excisional biopsy or organ-sparing procedures such as debulking of airway-compromising tumors. Residual measurable tumor is required for enrollment as discussed above.
10. Participants receiving other investigational agents.
11. Prior systemic anti-cancer treatment within the last 8 weeks.
12. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer or any tumors that are not likely to influence life expectancy in the subsequent 3 years without active treatment.
13. Has known history of, or any evidence of active, non-infectious pneumonitis.
14. Has known active Hepatitis B or hepatitis C. If eradicated, patient is eligible.
15. Has received a live vaccine within 28 days of planned start of study therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2024-07-17 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1 Primary Outcome: Phase 1 Dose of HB-201 and HB-201/202 Combined with Chemotherapy | 2 years
  The phase 1 dose of HB-201 monotherapy and alternating HB-201 and 202 therapy in combination with chemotherapy in patients with HPV 16 head and neck cancer as assessed by data on reported dose-limiting toxicities (side effects) among participants. These side effects will be measures according to the Common Terminology Criteria for Adverse Events version 5
Phase 2 Primary Outcome: Deep Response Rate of Participants Treated with HB-201 or HB-201/202 Combined with Chemotherapy | 2 years
  The deep response rate (DRR) of participants who receive neoadjuvant HB-201 monotherapy combined with chemotherapy or alternating doses of HB-201 and HB-202 combined with chemotherapy. This response rate will be assessed by tumor shrinkage according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
Correlation Between Plasma HPV-DNA and Tumor HPV-DNA | 2 years
  Correlation between plasma HPV-DNA and tumor HPV-DNA as assessed by an analysis of plasma and sputum samples of participants using next generation sequencing analysis.
Changes in Plasma HPV-DNA During Study Treatment with HB-201 and Alternating HB201/202 Combined with Chemotherapy | 2 years
  Changes in the amount of HPV-DNA found in plasma during neoadjuvant HB-201 monotherapy and HB-201 and HB-202 alternating two-vector therapy combined with chemotherapy as assessed by next generation sequencing analysis of participants' plasma samples.
Pathologic Response in Participants Undergoing Transoral Robotic Surgery (TORS) | 2 years
  Pathologic response in patients undergoing TORS following neoadjuvant HB-201 monotherapy and HB-202 alternating two-vector therapy combined with chemotherapy. Response will be assessed by tumor shrinkage according to Response Evaluation Criteria in Solid Tumors 1.1.
Progression Free Survival | 2 years
  Progression-free survival of participants as assessed by data recorded in study/clinical records and statistical analysis.
Overall Survival | 2 years
  Overall survival of participants as assessed by data recorded in study/clinical records and statistical analysis.
Locoregional Control | 2 years
  Locoregional control of participants as assessed by data recorded in study/clinical records and statistical analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ari Rosenberg, MD, Principal Investigator — University of Chicago - Comprehensive Cancer Center
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes